CLINICAL TRIAL: NCT04885179
Title: Sphingosine Phosphate Lyase Insufficiency Syndrome - Observational Study and Patient Registry (International)
Brief Title: SPL Insufficiency Syndrome (SPLIS)/NPHS14: a SPLIS Observational Study and Patient Registry (International)
Acronym: SPLIS-OSPRI
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20-32291
Record Dates: First submitted 2021-04-29; First posted 2021-05-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Sphingolipidoses; Enzyme Deficiency
Keywords: SPLIS; sphingosine phosphate lyase; SGPL1; sphingolipidosis; steroid-resistant nephrotic syndrome; primary adrenal insufficiency; neurological defect
MeSH Terms: conditions — Sphingolipidoses; Nephrotic Syndrome; Addison Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Leftover skin biopsy material or fibroblasts derived from skin biopsies obtained as part of medical care may be used to create a cell line that will be analyzed and stored in a SPLIS specimen bank at UCSF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with SPLIS: Individuals diagnosed with SPLIS based on genetic testing that confirms bi-allelic pathogenic variants in SGPL1
  Interventions: Other: no intervention
- Parents of individuals with SPLIS: Parents of individuals diagnosed with SPLIS based on genetic testing that confirms bi-allelic pathogenic variants in SGPL1
  Interventions: Other: no intervention
- age and gender-matched controls: The investigators will attempt to collect biological specimens from individuals closely matched to SPLIS patient cohort by age and gender. This group may include siblings, cousins, and unrelated healthy children and adults.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No interventions are involved in this observational study.

SUMMARY:
This protocol aims to gather information about sphingosine phosphate lyase insufficiency syndrome (SPLIS), also known as NPHS14, and to create a SPLIS patient registry. Medical records, radiological and pathology results, blood test results, and genetic information will be collected. Samples of blood, cheek cells, urine and stool may be collected for analysis. If a skin biopsy has been performed for medical care, cells from the biopsy may be analyzed. No treatment or other intervention is involved in this study. However, the effect of treatments administered by the patient's physician may be detected and monitored based on changes in the blood or urine.

DETAILED DESCRIPTION:
This protocol aims to gather information about sphingosine phosphate lyase insufficiency syndrome (SPLIS), a condition also known as NPHS14 or familial steroid-resistant nephrotic syndrome with adrenal insufficiency. SPLIS is a recently discovered genetic disease caused by recessive mutations in the SGPL1 gene. SPLIS can have effects on the kidney, adrenal gland, brain, skin, and blood cells. Some patients with SPLIS do not survive beyond infancy, whereas others live to adulthood. By monitoring the natural history of SPLIS over time in affected patients, the investigators will establish a clinical baseline that reflects how the disease progresses over time. This information may be useful in future clinical trials. The results may reveal which types of SGPL1 mutations correlate with best and worst patient outcomes. Some SPLIS patients are current on a regimen of high dose vitamin B6 supplementation on the advice of their treating physician. By including patients treated with B6, our study may provide evidence for the impact of B6 treatment on biochemical and blood markers of the disease. Our overall goals are to characterize the clinical, biochemical and metabolic manifestations of SPLIS and how these manifestations change over time within individuals with this condition.

ELIGIBILITY:
Inclusion Criteria: Individuals of all ages diagnosed with SPLIS based on bi-allelic pathogenic variants of SGPL1, including children and neonates, as well as family members or caregivers, healthy volunteers and individuals with other sphingolipidoses.

Exclusion Criteria: the investigators will not include:

* prisoners
* pregnant women
* healthy volunteers with:

  * diabetes,
  * infection,
  * fever,
  * known HIV/AIDS,
  * cardiac disease
  * or anemia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SPLIS is a genetic disorder caused by recessive mutations in SGPL1. The study population includes individuals with confirmed bi-allelic mutations in SGPL1, regardless of age, gender, disease manifestations, or treatments received. Some patients with SPLIS will have kidney failure, adrenal insufficiency and/or neurological problems. Parents, family members and unrelated healthy individuals enrolled during routine health appointments, elective surgical procedures and other medical interactions will be included as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival | 0-99 years
  The primary outcome of this study is survival (age at death).

SECONDARY OUTCOMES:
Onset of nephrotic syndrome | 0-99 years
  Age at onset of proteinuria greater than 3.5 grams per 24h

OTHER OUTCOMES:
Onset of primary adrenal insufficiency | 0-99 years
  Age at onset of glucocorticoid insufficiency with or without other endocrine defects
Responsiveness of blood sphingolipid levels to vitamin B6 supplementation | 0-99 years
  Changes in blood sphingolipid levels before and after caring physician-initiated vitamin B6 supplementation
Skin fibroblast sphingolipid levels in response to vitamin B6 | 1-6 weeks
  Skin fibroblast sphingolipid levels compared by liquid chromatography/mass spectrometry in medium containing various forms of vitamin B6 or lacking vitamin B6.
Responsiveness of absolute lymphocyte count to vitamin B6 supplementation | 0-99 years
  Changes in blood absolute lymphocyte count before and after caring physician-initiated vitamin B6

CONTACTS AND LOCATIONS:
Overall Officials: Julie D Saba, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lovric S, Goncalves S, Gee HY, Oskouian B, Srinivas H, Choi WI, Shril S, Ashraf S, Tan W, Rao J, Airik M, Schapiro D, Braun DA, Sadowski CE, Widmeier E, Jobst-Schwan T, Schmidt JM, Girik V, Capitani G, Suh JH, Lachaussee N, Arrondel C, Patat J, Gribouval O, Furlano M, Boyer O, Schmitt A, Vuiblet V, Hashmi S, Wilcken R, Bernier FP, Innes AM, Parboosingh JS, Lamont RE, Midgley JP, Wright N, Majewski J, Zenker M, Schaefer F, Kuss N, Greil J, Giese T, Schwarz K, Catheline V, Schanze D, Franke I, Sznajer Y, Truant AS, Adams B, Desir J, Biemann R, Pei Y, Ars E, Lloberas N, Madrid A, Dharnidharka VR, Connolly AM, Willing MC, Cooper MA, Lifton RP, Simons M, Riezman H, Antignac C, Saba JD, Hildebrandt F. Mutations in sphingosine-1-phosphate lyase cause nephrosis with ichthyosis and adrenal insufficiency. J Clin Invest. 2017 Mar 1;127(3):912-928. doi: 10.1172/JCI89626. Epub 2017 Feb 6. PMID 28165339
- [Background] Prasad R, Hadjidemetriou I, Maharaj A, Meimaridou E, Buonocore F, Saleem M, Hurcombe J, Bierzynska A, Barbagelata E, Bergada I, Cassinelli H, Das U, Krone R, Hacihamdioglu B, Sari E, Yesilkaya E, Storr HL, Clemente M, Fernandez-Cancio M, Camats N, Ram N, Achermann JC, Van Veldhoven PP, Guasti L, Braslavsky D, Guran T, Metherell LA. Sphingosine-1-phosphate lyase mutations cause primary adrenal insufficiency and steroid-resistant nephrotic syndrome. J Clin Invest. 2017 Mar 1;127(3):942-953. doi: 10.1172/JCI90171. Epub 2017 Feb 6. PMID 28165343
- [Background] Weaver KN, Sullivan B, Hildebrandt F, Strober J, Cooper M, Prasad R, Saba J. Sphingosine Phosphate Lyase Insufficiency Syndrome. 2020 Oct 15. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK562988/ PMID 33074640
- [Background] Choi YJ, Saba JD. Sphingosine phosphate lyase insufficiency syndrome (SPLIS): A novel inborn error of sphingolipid metabolism. Adv Biol Regul. 2019 Jan;71:128-140. doi: 10.1016/j.jbior.2018.09.004. Epub 2018 Sep 25. PMID 30274713
- [Background] Zhao P, Liu ID, Hodgin JB, Benke PI, Selva J, Torta F, Wenk MR, Endrizzi JA, West O, Ou W, Tang E, Goh DL, Tay SK, Yap HK, Loh A, Weaver N, Sullivan B, Larson A, Cooper MA, Alhasan K, Alangari AA, Salim S, Gumus E, Chen K, Zenker M, Hildebrandt F, Saba JD. Responsiveness of sphingosine phosphate lyase insufficiency syndrome to vitamin B6 cofactor supplementation. J Inherit Metab Dis. 2020 Sep;43(5):1131-1142. doi: 10.1002/jimd.12238. Epub 2020 May 4. PMID 32233035
- [Background] Martin KW, Weaver N, Alhasan K, Gumus E, Sullivan BR, Zenker M, Hildebrandt F, Saba JD. MRI Spectrum of Brain Involvement in Sphingosine-1-Phosphate Lyase Insufficiency Syndrome. AJNR Am J Neuroradiol. 2020 Oct;41(10):1943-1948. doi: 10.3174/ajnr.A6746. Epub 2020 Aug 27. PMID 32855188
- [Background] Zhao P, Tassew GB, Lee JY, Oskouian B, Munoz DP, Hodgin JB, Watson GL, Tang F, Wang JY, Luo J, Yang Y, King S, Krauss RM, Keller N, Saba JD. Efficacy of AAV9-mediated SGPL1 gene transfer in a mouse model of S1P lyase insufficiency syndrome. JCI Insight. 2021 Apr 22;6(8):e145936. doi: 10.1172/jci.insight.145936. PMID 33755599